CLINICAL TRIAL: NCT04550676
Title: High-Intensity Exercise to Attenuate Limitations and Train Habits in Older Adults With HIV
Acronym: HEALTH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Case Western Reserve University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-1985
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Hiv; Fatigue; Mobility Limitation
Keywords: mitochondrial function; physical function; frailty; exercise
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Fatigue; Mobility Limitation; Frailty; Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants will first be randomized to continuous moderate intensity or high-intensity interval training for 16 weeks. After 16 weeks, participants will be re-randomized to 12-week coaching intervention or control.
Masking Description: Outcomes assessors will be blinded for endpoints, as feasible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (Experimental)
  Interventions: Behavioral: HIIT (intervention)
- Continuous moderate intensity exercise (Active Comparator)
  Interventions: Behavioral: CME (active control)

INTERVENTIONS:
Behavioral: HIIT (intervention) — Following a 5-minute warm-up, high and moderate-intensity exercise bouts will alternate: a five bouts of 4-minute high-intensity exercise (90% VO2peak) will alternate with four 3-minute bouts of moderate-intensity exercise (50% VO2peak) by week 8. This is followed by a 5-minute cool-down. The total exercise time will be 42 minutes. For resistance exercise, the initial goal will be to complete 3 sets of 8-10 repetitions of 3 exercises at low intensity (50% 1-RM) and then progress to moderate intensity (70-80% 1-RM). Exercise intensity will increase every 4 weeks or when participants can complete more than 8 repetitions with proper form at the prescribed weight.
  Arms: High intensity interval training
Behavioral: CME (active control) — Following a 4-minute warm-up, the participant will walk/jog for up to 42 continuous minutes at 60% VO2peak. This is followed by a 4-minute cool-down. The total exercise time is 50 minutes. For resistance exercise, the initial goal will be to complete 3 sets of 8-10 repetitions of 3 exercises at low intensity (50% 1-RM) and then progress to moderate intensity (70-80% 1-RM). Exercise intensity will increase every 4 weeks or when participants can complete more than 8 repetitions with proper form at the prescribed weight.
  Arms: Continuous moderate intensity exercise

SUMMARY:
This is a multi-site, randomized, single-blind (researchers), active treatment concurrent control trial with individuals aged 50-80 living with HIV who experience fatigue and live a sedentary lifestyle. The overall goals of this proposal are to determine whether high-intensity interval training (HIIT) can overcome physical function impairments and increased fatigue (Aim 1) and impairments in mitochondrial bioenergetics of older people with HIV (PWH) to a greater extent than continuous moderate-intensity exercise (CME) (Aim 2). The investigators further seek to determine whether a biobehavioral coaching intervention following either HIIT or CME can promote long-term adherence to physical activity (Aim 3), a crucial component of the sustainability of the intervention. This study will enroll 100 participants in Aurora, Colorado and Seattle, Washington. Data collection will occur at each visit, with baseline data collected at the initial visit. A 3-month follow-up will be conducted over the phone from the date of the final visit.

The initial enrollment goal of 100 was increased to 120 in 2023 to facilitate a larger number of participants with key secondary outcomes.

DETAILED DESCRIPTION:
This is a multi-site, randomized, single-blind (researchers), active treatment concurrent control trial with individuals aged 50 and older living with HIV who experience fatigue and live a sedentary lifestyle. The overall goals of this proposal are to determine whether high-intensity interval training (HIIT) can overcome physical function impairments and increased fatigue (Aim 1) and impairments in mitochondrial bioenergetics of older people with HIV (PWH) to a greater extent than continuous moderate-intensity exercise (CME) (Aim 2). The investigators further seek to determine whether a biobehavioral coaching intervention following either HIIT or CME can promote long-term adherence to physical activity (Aim 3), a crucial component of the sustainability of the intervention. This study will enroll 100 participants in Aurora, Colorado and Seattle Washington.

Physical function will be measured by a 400-meter walk test (400MWT) and the short physical performance battery in its original (SPPB) and modified (mSPPB) forms. Fatigue will be measured by the Lee Fatigue Scale (LFS) - a 7-item visual analog self-report scale that asks participants to rate from 0 to 10 how they feel "right now." Mitochondrial bioenergetics will be assessed through blood draws, muscle biopsies and mitochondrial assays. Adherence to physical activity (PA) will be analyzed through ActiGraphy - measurement of PA duration and intensity on three planes of movement captured through PA monitors.

Finally, perceptions of PA will be determined through the analysis of qualitative interviews.

The hypotheses are that that investigators will see greater changes in mitochondrial bioenergetics with HIIT (AIM 1), and that these changes will be related to improved physical function and fatigue (Aim 2). The investigators expect that HIIT will result in greater exercise satisfaction and likelihood of long-term continuation of exercise (Aim 3). Using a coaching intervention for self-directed exercise that combines motivational interviewing and personalized support during the maintenance phase (Aim 3), the investigators seek to develop the ideal "cocktail" to promote healthspan among older PWH in the current era of ART.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 50years,
* Sedentary lifestyle, defined by self-reported physical activity that breaks a sweat <3 days/week, with no regular resistance exercise for 3 months preceding study,
* Fatigued (≥2.0 on either of the first two screening items on the HIV-Related Fatigue Scale),
* HIV infection, on prescribed HIV antiretroviral therapy for ≥ 12 months, with no current use (within 1 year) of older drugs with established mitochondrial toxicity (i.e., D4T, DDI, ZDV),
* HIV-1 RNA level < 200 copies/mL, for a minimum of 12 months prior to enrollment, with an allowed blip to 500 copies/mL presuming repeat assessments are below 200 copies,
* Willing to participate in either assigned arm of a 16-week supervised exercise intervention 3 times weekly,
* Thyroid Stimulating Hormone (TSH) within normal lab limits-Cell phone with ability to receive text messaging in order to participate in the biobehavioral maintenance intervention or ability to access to email daily
* Ability and willingness of participant to provide informed consent and consent for access to medical record
* COVID-19 vaccination and appropriate boosters received

Exclusion Criteria:

* Weight over 450 pounds (due to limitations of the DXA machine)
* Use of sex hormone therapy, if on for ≤3 months (stable doses for >3 months will be permitted)
* Use of other hormone replacement, if on for ≤ 3 months (stable doses >3 months will be permitted)
* Anemia (Hemoglobin ≤9 g/dL for women or ≤10 g/dL for men) due to contribution to fatigue,
* Diagnosis of mitochondrial disease For participants undergoing the muscle biopsy only, use of anticoagulant therapy other than low dose aspirin that cannot be held for at least 7 days for the muscle biopsy. Aspirin and non-steroidal use will be permitted but will be held for 7 days prior to the muscle biopsy, and can be resumed following the biopsy.
* Due to the expected fatigue associated with COVID-19 and potential infection risk, anyone with a diagnosis of COVID will not be eligible for enrollment until at least 30 days after symptom resolution and return to baseline level of function.
* Active substance abuse or other factors that could prevent compliance or safety with study visits, at the discretion of the site investigator,
* Reasons for medical exclusion, as determined by study PIs:
* Uncontrolled hypertension defined as resting systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg; participants who do not meet these criteria at first screening will be re-evaluated, including follow-up evaluation by their primary care provider with initiation or adjustment of anti-hypertensive medications,
* Unstable ischemic heart disease (e.g., angina, ST segment depression) or serious arrhythmias at rest or during the graded exercise test without negative follow-up evaluation will be cause for exclusion; follow-up evaluation must include diagnostic testing (e.g., thallium stress test) with interpretation by a cardiologist,
* New York Heart Association Class III or IV congestive heart failure, clinically significant aortic stenosis, uncontrolled angina, or uncontrolled arrhythmia,
* Pulmonary disease requiring the use of supplemental oxygen at rest or with physical exertion,
* Malignancy requiring chemotherapy or radiation therapy within 24 weeks prior to enrollment,
* Poorly controlled diabetes, as evidenced by hemoglobin A1c > 8.0, documented within 6 months of study visit,
* Surgery/trauma/injury/fracture within 24 weeks prior to enrollment that, in the opinion of the study physician, may impact a subject's baseline functional testing and ability to exercise,
* Balance impairments that may impact functional testing and ability to safely exercise as reported by the participant or in their medical record,
* Orthopedic problems (e.g., severe osteoarthritis, rheumatoid arthritis) that greatly limit the ability to perform moderate intensity resistance exercise (e.g., unable to be properly positioned in exercise equipment or to have severely restricted range of motion even after modifications have been made),
* Persons who, in the judgment of the study physician, appear to have unstable health or are incapable of safely participating in the exercise intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Any genders can be included
Enrollment: 118 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
Change in physical function | 0-16 weeks
  400-m walk time is a continuous measure of the total time required to complete a 400-m walking course. Lower values indicate a faster walking speed.

SECONDARY OUTCOMES:
Change in fatigue | 0-16 weeks
  The Lee Fatigue Score measures severity of fatigue. Possible scores range from 0 to 10, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Erlandson, MD, Principal Investigator — University of Colorado, Denver; Allison Webel, PhD, RN, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - University of Colorado - Anschutz Medical Campus, Aurora, Colorado
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set may be shared with investigators upon written request, review and approval by institutional officials, and establishing a data use agreement. Investigators requesting other study documents (protocol, analysis plan, informed consent, code, etc) should contact the study team.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The investigators will make the following available upon request after the primary manuscript is published: the trial description information, protocol, SAP, ICF. Data will be posted to ClinicalTrials.gov after publication of the primary manuscript. Until that time, a message will also appear stating that the trial data will be available after publication of the primary manuscript.
Access Criteria: Investigators interested in acquiring study data should contact the study team. Sharing of de-identified data will be considered upon review/approval of the request by the Institutional Review Board, with a data use agreement.

REFERENCES:
- [Background] Oliveira VHF, Erlandson KM, Cook PF, Jankowski C, MaWhinney S, Dirajlal-Fargo S, Knaub L, Hsiao CP, Horvat Davey C, Webel AR. The High-Intensity Exercise Study to Attenuate Limitations and Train Habits in Older Adults With HIV (HEALTH): A Research Protocol. J Assoc Nurses AIDS Care. 2022 Mar-Apr 01;33(2):178-188. doi: 10.1097/JNC.0000000000000276. PMID 34039876